CLINICAL TRIAL: NCT07105592
Title: A Prospective, Phase Ib/II Study of Nimotuzumab Combined With Adebrelimab and Chemotherapy for the Treatment of Patients With Recurrent/Metastatic Head And Neck Squamous Cell Carcinoma Who Are Ineligible to High-Dose Cisplatin
Brief Title: A Study of Nimotuzumab Plus Adebrelimab With Chemotherapy in Cisplatin-Ineligible Patients With Head And Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ji Dongmei, Associate Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUSCC-HN-002
Record Dates: First submitted 2025-05-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: PD-L1 inhibitor; Nimotuzumab; Adebrelimab; Cisplatin intolerance; EGFR inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab+Adebrelimab+Chemotherapy (Experimental): Phase Ib Treatment Regimen:
  Nimotuzumab: Three dose groups (200 mg, 400 mg, 600 mg), administered via intravenous infusion over at least 60 minutes, once every 3 weeks, until disease progression, intolerable toxicity, or subject withdrawal from the trial.
  Adebrelimab: Fixed dose of 1200 mg, administered via intravenous infusion, once every 3 weeks, until disease progression, intolerable toxicity, or subject withdrawal from the trial.
  Albumin-bound Paclitaxel: 100 mg/m², administered intravenously on Days 1 and 8, once every 3 weeks, for 6 cycles.
  Carboplatin: AUC=2 (calculated using the Calvert formula), administered intravenously on Days 1 and 8, once every 3 weeks, for 6 cycles.
  Phase II Treatment Regimen:
  Nimotuzumab: Recommended Phase II dose (RP2D) as determined from Phase Ib, administered via intravenous infusion on Day 1, once every 3 weeks, until disease progression, intolerable toxicity, or subject withdrawal from the trial.
  Adebrelimab: Fixed dose of 1200 mg, administered vi
  Interventions: Drug: Nimotuzumab+Adebrelimab+Chemotherapy

INTERVENTIONS:
Drug: Nimotuzumab+Adebrelimab+Chemotherapy — Phase Ib Treatment Regimen:
  Nimotuzumab: Three dose groups (200 mg, 400 mg, 600 mg), administered via intravenous infusion over at least 60 minutes, once every 3 weeks, until disease progression, intolerable toxicity, or subject withdrawal from the trial.
  Adebrelimab: Fixed dose of 1200 mg, administered via intravenous infusion, once every 3 weeks, until disease progression, intolerable toxicity, or subject withdrawal from the trial.
  Albumin-bound Paclitaxel: 100 mg/m², administered intravenously on Days 1 and 8, once every 3 weeks, for 6 cycles.
  Carboplatin: AUC=2 (calculated using the Calvert formula), administered intravenously on Days 1 and 8, once every 3 weeks, for 6 cycles.
  Phase II Treatment Regimen:
  Nimotuzumab: Recommended Phase II dose (RP2D) as determined from Phase Ib, administered via intravenous infusion on Day 1, once every 3 weeks, until disease progression, intolerable toxicity, or subject withdrawal from the trial.
  Adebrelimab: Fixed dose of 1200 mg, administered via

SUMMARY:
This is a prospective, single-arm, Phase Ib/II clinical study to evaluate the safety and efficacy of nimotuzumab combined with adebrelimab and chemotherapy in patients with recurrent and metastatic head and neck squamous cell carcinoma who are ineligible to high-dose cisplatin treatment.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, Phase Ib/II clinical trial. Phase Ib uses a 3+3 dose escalation design, and Phase II uses a Simon two-stage design. Phase Ib explores the proper dosage of nimotuzumab to combine with adebrelimab and chemotherapy in patients with recurrent and metastatic head and neck squamous cell carcinoma who are ineligible to high-dose cisplatin treatment. Phase II explores the efficacy and safety of nimotuzumab combined with adebrelimab and chemotherapy in the same patient population. It is expected to enroll approximately 68 subjects with recurrent and metastatic head and neck squamous cell carcinoma who are ineligible to high-dose cisplatin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years.
2. Diagnosis: Histologically or cytologically confirmed recurrent or metastatic head and neck squamous cell carcinoma, meeting the following conditions:Local treatment methods cannot achieve a cure (including cases where the patient refuses local treatment or is deemed unsuitable for local treatment by the physician, e.g., inability to tolerate anesthesia or other factors precluding local radiotherapy).No prior systemic treatment (targeted therapy, immunotherapy, and/or chemotherapy) after recurrence or metastasis.Primary nasopharyngeal carcinoma is not permitted.
3. Cisplatin Intolerance: Patients must have at least one of the following reasons for being unsuitable for cisplatin-based chemotherapy:Age >70 years.Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 2.Renal function impairment (creatinine clearance <50 mL/min). If this criterion is met, the creatinine clearance standard in criterion 7 is not applicable.Severe tinnitus or hearing loss (requiring a hearing aid or showing a ≥25 dB shift at two consecutive frequencies on audiometry).Inability to receive intravenous hydration due to cardiac dysfunction or other comorbidities (left ventricular ejection fraction [LVEF] <50%).Patient refusal of cisplatin-based chemotherapy.
4. Oropharyngeal Cancer: Availability of tumor tissue for P16/HPV testing (if previously tested, retesting is not required).
5. Performance Status: ECOG PS score of 0-2.
6. Measurable Disease: At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
7. Adequate organ function：Hematology:Absolute Neutrophil Count (ANC): ≥1500/μL (1.5 × 10⁹/L),Platelets: ≥100,000/μL (100 × 10⁹/L),Hemoglobin: ≥9 g/dL (90 g/L) or ≥5.6 mmol/L.Renal:Serum Creatinine or Creatinine Clearance: Creatinine ≤1.5 × Upper Limit of Normal (ULN); if creatinine >1.5 × ULN, then creatinine clearance must be ≥60 mL/min.Hepatic:Total Bilirubin: ≤1.5 × ULN,Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT): ≤2.5 × ULN; if liver metastases are present, then ≤5 × ULN.Coagulation:International Normalized Ratio (INR) or Prothrombin Time (PT): ≤1.5 × ULN; if the patient is receiving anticoagulant therapy, PT or Partial Thromboplastin Time (PTT) must be within the therapeutic range for the anticoagulant used.
8. PD-L1 Testing: Availability of tumor tissue (from the tumor core or resected tumor) for PD-L1 testing (if previously tested, additional testing is not required).
9. Reproductive Status:Female subjects must have a negative pregnancy test within two weeks before starting study treatment and must not be breastfeeding.Female subjects must agree to use effective contraception during the study and for 6 months after the last dose of study drug.Male subjects must agree to use effective contraception during the study and for 6 months after the last dose of study drug.
10. Informed Consent: Subjects must voluntarily participate in the study, provide written informed consent, and be able to comply with the protocol-specified visits and procedures.

Exclusion Criteria:

1. Curable by Local Treatment: Patients whose disease can be cured by local treatment methods. Exceptions include cases where the patient refuses local treatment or is deemed unsuitable for local treatment by the investigator (specific reasons must be documented at enrollment).
2. Recent Local Treatment or Unresolved Adverse Events: Patients who have undergone radiotherapy or other local treatments (e.g., surgery) within 2 weeks prior to enrollment, or who have not recovered from adverse events (AEs) from prior treatments (i.e., AEs ≤ Grade 1 or returned to baseline). Exceptions include:Peripheral neuropathy ≤ Grade 2. Alopecia ≤ Grade 2.Laboratory abnormalities meeting inclusion criterion 7 (adequate organ function).
3. Recent Clinical Trial Participation: Patients who participated in another clinical trial within 4 weeks prior to enrollment (except those in the follow-up period who did not receive treatment).
4. Poor Prognosis: Patients with an estimated life expectancy of less than 3 months as assessed by the investigator, or those with rapidly progressing disease (e.g., tumor bleeding or uncontrolled tumor pain).
5. Immunosuppression: Patients diagnosed with an immunodeficiency disease within 7 days prior to enrollment, or those receiving systemic corticosteroid therapy or other immunosuppressive treatments. Exceptions include:Use of contrast agents.Corticosteroid use for managing AEs.Physiological doses of corticosteroids as determined by the investigator.
6. Other Malignancies: Patients diagnosed with another malignant tumor within 5 years prior to enrollment. Exceptions include:Cured basal cell carcinoma of the skin.Cured squamous cell carcinoma of the skin.Cervical carcinoma in situ.Breast carcinoma in situ.Other cured tumors deemed acceptable by the investigator.
7. Active CNS Metastases: Patients with known active central nervous system (CNS) metastases. Exceptions include patients with stable CNS metastases for at least 4 weeks prior to enrollment (confirmed by stable CT or MRI, no new lesions, no progression of existing lesions, resolution of neurological symptoms to baseline, and no corticosteroid use for at least 7 days). Patients with carcinomatous meningitis, regardless of stability, are excluded.
8. Active Autoimmune Disease: Patients with an active autoimmune disease requiring systemic treatment within 2 years prior to enrollment (e.g., disease-modifying agents, corticosteroids, or immunosuppressants). Exceptions include replacement therapies (e.g., thyroxine, insulin, or physiological doses of corticosteroids for adrenal or pituitary insufficiency).
9. Organ or Tissue Transplantation: Patients who have received allogeneic tissue or solid organ transplantation.
10. Non-Infectious Pneumonitis: Patients with a history of non-infectious pneumonitis requiring corticosteroid treatment or current pneumonitis.
11. Active Infection: Patients with an active infection requiring systemic treatment.
12. Other Safety Concerns: Patients with medical conditions or histories that, in the investigator's judgment, may compromise safety or interfere with study assessments.
13. Mental Health or Substance Abuse: Patients with psychiatric disorders or substance abuse issues that may affect study compliance or cooperation.
14. Pregnancy or Reproductive Plans: Pregnant or breastfeeding women, or individuals planning to conceive from the start of the screening period until 180 days after the last dose of study drug.
15. HIV Infection: Patients with positive HIV serology or a history of HIV infection.
16. Active Hepatitis: Patients with active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
17. Recent Live Vaccine: Patients who received a live vaccine within 30 days prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Phase Ib:Dose-limiting toxicity (DLT) | 3 weeks after treatment initiation
  Occurrence of specific severe toxicities (grade 3 or 4) related to the treatment during the first cycle.
Phase II:Objective response rate (ORR) | 2 years after enrollment of final patient
  Objective response rate measured as number of complete and partial response divided by the number of patients included.

SECONDARY OUTCOMES:
Phase Ib:Objective response rate (ORR) | 2 years after enrollment of final patient
  Objective response rate measured as number of complete and partial response divided by the number of patients included.
Phase Ib/Phase II::Disease control rate (DCR) | 2 years after enrollment of final patient
  Disease control rate measured as number of complete and partial response or stable disease divided by the number of patients included.
Phase Ib/Phase II:Progression-free Survival (PFS) | up to 2 years
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Phase Ib/Phase II:Overall Survival (OS) | up to 2 years
  Overall Survival (OS) (median) was determined using the number of months measured from the initial date of treatment to the recorded date of death of participants.
Phase II:Safety | Since the signing of informed consent forms to 30 days after the last cycle
  Incidence of Treatment-Emergent Adverse Events (CTCAE 5.0）
Phase II:Quality of life | up to 2 years
  Assessed using EORTC QLQ-C30 (V3) questionnaires.The EORTC QLQ-C30 is a 30-item validated questionnaire designed to assess the quality of life in cancer patients. It includes five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea/vomiting), a global health status/quality of life scale, and six single items assessing additional symptoms (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All scales and single items are scored on a range from 0 to 100. For the functional scales and global health status scale, higher scores indicate better quality of life or functioning. For the symptom scales and single items, higher scores indicate worse symptoms or greater severity.
Phase II:Quality of life | up to 2 years
  Assessed using EORTC QLQ-H&N35 questionnaires.The EORTC QLQ-H&N35 is a 35-item validated questionnaire specifically designed to assess quality of life in head and neck cancer patients. It includes seven symptom scales (pain, swallowing, senses, speech, social eating, social contact, and sexuality) and eleven single items addressing additional head and neck-specific symptoms (e.g., teeth problems, mouth opening, dry mouth, sticky saliva, coughing, feeling ill, use of painkillers, nutritional supplements, feeding tube, weight loss, and weight gain). All scales and single items are scored on a range from 0 to 100, with higher scores indicating worse symptoms or greater severity.
Phase II:Impact of tumor-related biomarkers on prognosis | 2 years after enrollment of final patient
  Analysis of how specific biomarkers correlate with patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dongmei Ji, doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No